CLINICAL TRIAL: NCT06919380
Title: Safety and Efficacy Study of Nebulized Mesenchymal Stem Cell-Derived Exosomes (MSC-exos) for the Treatment of Anti-MDA5 Positive Dermatomyositis-Associated Rapidly Progressive Interstitial Lung Disease (RP-ILD)
Brief Title: Nebulized MSC-Exos for Anti-MDA5+ RP-ILD: Safety and Efficacy Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Li Shiyue (Other)
Responsible Party: Sponsor-Investigator, Li Shiyue, professor, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2024 -156 -01
Record Dates: First submitted 2025-02-13; First posted 2025-04-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Anti-MDA5 Positive Dermatomyositis-Associated RP-ILD; Rapidly Progressive Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Anti-MDA5 Positive; Rapidly Progressive Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nebulized MSC-exos for Anti-MDA5+ RP-ILD Treatment (Experimental): This arm of the study involves the administration of nebulized Mesenchymal Stem Cell-derived Exosomes (MSC-exos-P1) as an intervention for patients diagnosed with Anti-MDA5 Positive Dermatomyositis-Associated Rapidly Progressive Interstitial Lung Disease (RP-ILD).
  Interventions: Drug: MSC-exos Nebulization Therapy

INTERVENTIONS:
Drug: MSC-exos Nebulization Therapy — The intervention in this study, "Nebulized MSC-exos for Anti-MDA5+ RP-ILD Treatment," is distinguished by its use of mesenchymal stem cell-derived exosomes (MSC-exos) for direct pulmonary delivery via nebulization. This targeted approach aims to modulate immune responses and reduce inflammation specific to lung diseases, offering a novel therapeutic strategy. This method stands out for its potential to provide a safer and more effective treatment for RP-ILD compared to traditional therapies.

SUMMARY:
Objective: To assess the safety, tolerability, and efficacy of nebulized MSC-exos-P1 in patients with anti-MDA5 positive dermatomyositis-associated rapidly progressive interstitial lung disease (RP-ILD).

Design: Prospective interventional trial with 10 eligible patients aged 18-75, meeting criteria for RP-ILD and anti-MDA5 positivity. Primary endpoint is safety and tolerability, measured by adverse events within 30 days post-treatment. Secondary endpoints are clinical improvements on days 14 and 28, including serological indicators and chest HRCT scores.

Exclusions: Pregnant/breastfeeding individuals, severe allergies, active pulmonary infections, pulmonary embolism, extracorporeal support treatments, and other specified conditions.

Treatment: Nebulized MSC-exos-P1 daily for 14 days, plus standard care of corticosteroids and immunosuppressants.

Monitoring: Regular vital signs, oxygenation index, and pulmonary function tests. Follow-ups at multiple points up to 12 months.

DETAILED DESCRIPTION:
This single-center, prospective interventional trial aims to evaluate the safety profile and potential efficacy of nebulized mesenchymal stem cell-derived exosomes (MSC-exos-P1) in anti-MDA5 positive dermatomyositis patients with rapidly progressive interstitial lung disease. Anti-MDA5 positive RP-ILD represents a critical clinical challenge with mortality rates exceeding 50% despite aggressive immunosuppressive therapy, highlighting the urgent need for novel treatment approaches.

The trial will enroll 10 eligible patients who will receive a 14-day course of daily nebulized MSC-exos-P1 while continuing standard immunosuppressive therapy. Safety monitoring will include daily vital signs, laboratory tests, and adverse event documentation during the treatment period. Efficacy assessments will measure changes in oxygenation parameters, pulmonary function, inflammatory biomarkers, and CT imaging findings at days 14 and 28 compared to baseline.

The scientific rationale for this intervention is based on preclinical evidence demonstrating the immunomodulatory, anti-inflammatory, and anti-fibrotic properties of MSC-derived exosomes. These nanoparticles have shown the ability to modify alveolar macrophage phenotypes, reduce pro-inflammatory cytokine production, and suppress fibroblast activation - mechanisms that may directly target the pathophysiological processes driving RP-ILD in this patient population. The nebulized delivery system enables direct targeting of affected lung tissue while minimizing systemic exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion if they meet all of the following criteria:

  1. Positive for anti-MDA5 antibody dermatomyositis (according to the "Chinese Expert Consensus on the Diagnosis and Treatment of Anti-MDA5 Positive Dermatomyositis (2023 Edition)");
  2. Pulmonary lesions meet the diagnostic criteria for RP-ILD.

     Exclusion Criteria:
* Patients who meet any of the following criteria will be excluded from this study:

  1. Pregnant or breastfeeding women, or women planning pregnancy during the study, or men unwilling to use contraceptive measures throughout the trial period;
  2. History of severe allergies or allergies to the main active ingredients of the trial medication;
  3. Currently suffering from severe pulmonary infections, pneumothorax, or large pleural effusions;
  4. Currently diagnosed with pulmonary embolism;
  5. Currently undergoing mechanical ventilation through tracheal intubation;
  6. Currently undergoing extracorporeal life support treatments such as ECMO, CRRT, PMX-DHP, or plasma exchange;
  7. Currently suffering from severe heart failure, liver, or kidney insufficiency;
  8. Expected to undergo lung transplantation in the near future;
  9. Currently suffering from lung cancer or pulmonary nodules suspected to be early-stage lung cancer;
  10. Suffering from primary immunodeficiency diseases;
  11. Currently suffering from active infectious diseases, including but not limited to HIV positivity, active tuberculosis, etc., and deemed unsuitable for this trial by the researcher;
  12. Use of other trial medications within 28 days before starting treatment, which the researcher judges may interfere with the safety and efficacy assessment of this trial medication;
  13. Other situations deemed not in the best interest of the subject or unsuitable for participation in this study by the researcher, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Three-Month Mortality Rate and Safety of Nebulized MSC-exos P1 | 3 months post-treatment initiation]
  Mortality measured as the percentage of participants who died within three months post-treatment. Safety assessed by number and severity of adverse events using CTCAE v5.0.

SECONDARY OUTCOMES:
Oxygen Saturation | Baseline, day 14, and day 28 post-treatment initiation
  Oxygen Saturation: SpO2 (%) via pulse oximetry
CT Lesion Changes | Baseline, day 14, and day 28 post-treatment initiation
  CT Lesion Changes: Semi-quantitative scoring system (0-25)
Symptom Improvement | Baseline, day 14, and day 28 post-treatment initiation
  Symptom Improvement: VAS (0-10) for dyspnea and cough
C-reactive Protein (CRP) | Baseline, day 14, and day 28 post-treatment initiation
  Serum C-reactive Protein levels (CRP) (mg/L)
Interleukin-6 (IL-6) | Baseline, day 14, and day 28 post-treatment initiation
  Interleukin-6 (IL-6) (pg/mL)
D-dimer | Baseline, day 14, and day 28 post-treatment initiation
  Plasma D-dimer (μg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No